CLINICAL TRIAL: NCT03815149
Title: The Safety and Clinical Effectiveness of Pipeline™ Flex Embolization Devices With Shield Technology™ in Patients With Intracranial Aneurysms: a Multicentre Retrospective Study of an Australian Cohort (SCOPE-AUS)
Brief Title: Safety and Clinical Effectiveness of Pipeline™ Shield Devices for Intracranial Aneurysms
Acronym: SCOPE-AUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Prince of Wales Hospital, Sydney (Other Government); Liverpool Hospital, Sydney (Unknown); Sir Charles Gairdner Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GCMR0002; ISR-2017-10909 (Other Grant/Funding Number: Medtronic External Research Program)
Record Dates: First submitted 2018-10-06; First posted 2019-01-24 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Intracranial Aneurysm; Cerebral Aneurysm; Subarachnoid Hemorrhage; Stroke, Acute; Cerebral Hemorrhage; Cerebral Stroke; Neurologic Disorder
Keywords: Interventional Neuroradiology; Diagnostic neuroradiology; Neurosurgery; Neurovascular Devices; Flow Diversion Device
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Stroke; Cerebral Hemorrhage; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients with intracranial aneurysm(s): Standard of care elective, unscheduled or emergency procedures for the treatment of an unruptured or ruptured intracranial aneurysm(s) using a Pipeline™ Flex Embolization Device(s) with Shield Technology™
  Interventions: Device: Pipeline™ Flex Embolization Device with Shield Technology™

INTERVENTIONS:
Device: Pipeline™ Flex Embolization Device with Shield Technology™ — Neurointerventional procedures to treat intracranial (cerebral) aneurysms are minimally-invasive procedures performed by Interventional Neuroradiologists. The physician accesses the arterial system through a blood vessel in the groin followed by the insertion of a catheter. Pipeline™ Flex Embolization Device(s) with Shield Technology™,a flow diversion device, is implanted under high-magnification subtraction fluoroscopy, requiring the use of ancillary devices, such as micro-catheters and guidewires to complete the procedure under general anaesthetic. Procedural heparinisation and preloading with dual antiplatelet therapy (DAPT) using acetyl-salicylic acid and P2Y12 inhibitors such as clopidogrel or prasugrel are required.
  Other Names: Neurointerventional procedure

SUMMARY:
This observational, retrospective, single-arm, multi-centre cohort study will use real-world data (RWD) to develop real-world evidence (RWE) of the safety and clinical effectiveness of the Pipeline™ Flex Embolization Device with Shield Technology™ in Australian patients that have received a flow diversion device to treat an intracranial aneurysm (IA). The medical records from 500 procedures completed at Gold Coast University Hospital in Queensland (QLD), Prince of Wales Hospital in New South Wales (NSW), and Sir Charles Gardiner Hospital in Western Australia (WA), will be analysed.

The study will report the risk and likelihood of stroke (ischaemic and haemorrhagic), delayed neurological adverse events and incomplete aneurysm occlusion within sub-groups of the patient cohort and determine the predictive or confounding factors that influence clinical outcomes under pragmatic or 'real-world' conditions.

DETAILED DESCRIPTION:
Methodology summary: Single-arm, longitudinal, retrospective, multi-centre cohort study. A collaboration of Australian Interventional Neuroradiologists will create a data bank of existing clinical and angiographic data extracted from medical records review. The data collection variables are pre-specified using grading scales and clinical assessment with the greatest reliability or significant to to accurately represent patient cohorts receiving treatment within all indications of use. The study will establish a minimum dataset to collect patient socio-demographics, aneurysm characteristics, device characteristics, and clinical outcomes for up to 500 procedures completed using Pipeline™ Flex Embolization Device with Shield Technology™. A framework for data ab The prevalence, severity and outcomes of neurological adverse events of interest and bleeding events will be reported . Independent physician assessments of complete aneurysm occlusion from completed computed tomography scans (CT), Magnetic Resonance Imaging (MRI) scans and Digital Subtraction Angiography (DSA) procedures will be determined according to the Raymond Roy Occlusion Classification (MRRC), O'Kelly Marotta scale (OKM) for aneurysm occlusion using flow diverting devices and the Consensus grading scale for endovascular aneurysm occlusion up to 12 months post procedure. Assessments of wall apposition and in-stent stenosis (ISS) will also be completed.

Quality Assurance plan includes - Framework data abstraction - manual of procedures, data dictionary, data abstraction manual, desired inter-rater reliability +0.80; intrarater reliability, intraclass correlation coefficient (ICC) 0.75 - 0.9;

Medical imaging review assessed by assess aneurysm occlusion by an independent interventional neuroradiologist or a local physician operator that did not complete the primary procedure. Physician level of agreement - interrater reliability to be reported;

Independent physician review of all post-op strokes (ischaemic, haemorrhagic) cases to determine aetiology/mechanism;

Study personnel training; Site visits; remote data monitoring, data audits.

Statistical analysis plan include descriptive statistics and regression models to report prevalence, mortality, time-to-event analyses and estimations of risk; Counts of medical records with insufficient data for analysis or where the patient is identified as 'lost follow-up', this will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Medical records from patients that have received a Pipeline™ Flex Embolization Device with Shield Technology™ inclusive of all indications such as an elective procedure, unscheduled procedure or emergency procedure for an unruptured or ruptured intracranial aneurysm(s) at each study site
* Medical records from patients that have received other neurovascular therapies such as coils, intracranial stents etc. with a Pipeline™ Flex Embolization Device with Shield Technology™ used as an adjunctive device during the index procedure

Exclusion Criteria:

* Medical records from patients that have not received a Pipeline™ Flex Embolization Device with Shield Technology™ to treat an intracranial aneurysm

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is comprised of Australian patients aged ≥ 18 years that have received Pipeline™ Flex Embolization Devices with Shield Technology™ during a standard of care procedure to treat an IA. The patient selection period extends from 01 April 2015 to 30 June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stroke (short-term) | 30 days
  Prevalence and severity of ischaemic and haemorrhagic stroke post procedure
Mortality due to stroke (short-term) | 30 days
  Number of deaths due to ischaemic and haemorrhagic post procedure
Morbidity due to neurological adverse events of interest (short-term) | 30 days
  Prevalence of neurological adverse events of interest post procedure
Prevalence of stroke (long-term) | 12 months
  Prevalence and severity of ischaemic and haemorrhagic stroke post procedure
Morbidity due to neurological adverse events of interest (long-term) | 12 months
  Prevalence of neurological adverse events of interest post procedure
Mortality due to stroke (long-term) | 12 months
  Number of deaths due to ischaemic and haemorrhagic post procedure
Mortality due to neurological adverse events of interest (long-term) | 12 months
  Deaths due to other neurological adverse events of interest
All cause mortality | 12 months
  Deaths due to any cause

SECONDARY OUTCOMES:
Aneurysm occlusion - Wall apposition | Day 0
  Proportion of aneurysms with good wall apposition at post-operative time point
Aneurysm occlusion - Consensus grading scale for endovascular occlusion (short-term) | 6 months
  Proportion of aneurysms with Grade 0 - 5 aneurysm occlusion; Grade 0 is complete aneurysm occlusion (better outcome; maximum score) Grade 5 is less than 25% aneurysm occlusion (worse outcome; minimum score)
Aneurysm occlusion - Consensus grading scale for endovascular occlusion (long-term) | 12 months
  Proportion of aneurysms with Grade 0 - 5 aneurysm occlusion; Grade 0 is complete aneurysm occlusion (better outcome; maximum score) Grade 5 is less than 25% aneurysm occlusion (worse outcome; minimum score)
Aneurysm occlusion - O'Kelly Marotta Scale (OKM; short-term) | 6 months
  Proportion of aneurysms with Grade D1 aneurysm occlusion on the O'Kelly Marotta Scale. Grade D1 indicates completed aneurysms occlusion as seen on the arterial phase of the cerebral angiogram due to 0% filling (better outcome; maximum score). Grade A1 represents total filling of the aneurysm (>95%) as seen on the arterial phase of the cerebral angiogram (worse outcome; minimum score).
Aneurysm occlusion - O'Kelly Marotta Scale (OKM; long-term) | 12 months
  Proportion of aneurysms with Grade D1 aneurysm occlusion on the O'Kelly Marotta Scale; Grade D1 indicates completed aneurysms occlusion as seen on the arterial phase of the cerebral angiogram due 0% filling (better outcome; maximum score). Grade A1 represents total filling of the aneurysm (>95%) as seen on the arterial phase of the cerebral angiogram (worse outcome; minimum score).
Aneurysm occlusion - Modified Raymond Roy Classification (MRRC; short-term) | 6 months
  Proportion of aneurysms with Class 1 occlusion. Class 1 indicates complete obliteration of the aneurysm neck, representing complete aneurysm occlusion (better outcome; maximum score). Class 3b indicates residual aneurysm with contrast along aneurysm wall, representing substantial blood flow into the aneurysm, poor occlusion of aneurysm neck (worst outcome; minimum score).
Aneurysm occlusion - Modified Raymond Ray Classification (MRRC; long-term) | 12 months
  Proportion of aneurysms with Class 1 occlusion. Class 1 indicates complete obliteration of the aneurysm neck, representing complete aneurysm occlusion (better outcome; maximum score). Class 3b indicates residual aneurysm with contrast along aneurysm wall, representing substantial blood flow into the aneurysm, poor occlusion of aneurysm neck (worst outcome; minimum score).
Aneurysm occlusion - In-stent stenosis (ISS; short-term) | 30 days
  Proportion of aneurysms with Grade 2-4 ISS; ISS is a focal area of parent cerebral vessel narrowing caused by thrombosis or intimal hypoplasia. Grade 0 indicates no ISS is present (better outcome, maximum score). Grade 4 indicates occlusion of the cerebral parent vessel (worst outcome, minimum score).
Aneurysm occlusion - In-stent stenosis (ISS; short-term) | 90 days
  Proportion of aneurysms with Grade 2-4 ISS; ISS is a focal area of parent cerebral vessel narrowing caused by thrombosis or intimal hypoplasia.Grade 0 indicates no ISS is present (better outcome, maximum score). Grade 4 indicates occlusion of the cerebral parent vessel (worst outcome, minimum score).
Aneurysm occlusion - In-stent stenosis (ISS; long-term) | 6 months
  Proportion of aneurysms with Grade 2-4 ISS; ISS is a focal area of parent cerebral vessel narrowing caused by thrombosis or intimal hypoplasia.Grade 0 indicates no ISS is present (better outcome, maximum score). Grade 4 indicates occlusion of the cerebral parent vessel (worst outcome, minimum score).
Aneurysm occlusion - In-stent stenosis (ISS; long-term) | 12 months
  Proportion of aneurysms with Grade 2-4 ISS; ISS is a focal area of parent cerebral vessel narrowing caused by thrombosis or intimal hypoplasia.Grade 0 indicates no ISS is present (better outcome, maximum score). Grade 4 indicates occlusion of the cerebral parent vessel (worst outcome, minimum score).

OTHER OUTCOMES:
Functional outcomes - Modified Rankin Scale, nil disability | 90 days
  Change in mRS from baseline mRS 0-1; mRS is a clinician-reported measure of global disability. Level 0 indicates no disability (better outcome, maximum score). Level 6 indicates death (worst outcome, minimum score).
Functional outcomes - Modified Rankin Scale, disability | 90 days
  Change in mRS from baseline mRS 3-6; mRS is a clinician-reported measure of global disability. Level 0 indicates no disability (better outcome, maximum score). Level 5 indicates severe disability, bedridden, incontinent and requiring nursing care and attention (poor outcome, low score). Level 6 indicates death (worst outcome, minimum score).
Functional outcomes - number of days spent in hospital | 90 days
  mean time in hospital, an intensive care unit, or rehabilitation facility
Functional outcomes - home time post stroke | 90 days
  Number of days spent at home after a post-operative stroke
Procedural time | Day 0
  Time from start to end of the procedure
Dual anti platelet therapy (DAPT) - Assay values | Day 0
  % inhibition - DAPT assay values demonstrating impaired platelet activity
Bleeding events - The Bleeding Academic Research Consortium | 12 months
  Proportion, severity and classification of bleeding events
Re-treatment procedures | 12 months
  Proportion of aneurysms requiring re-treatment procedures
Incomplete aneurysms occlusion | 12 months
  Proportion of aneurysms with incomplete occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Henry (Hal) A Rice MBBS FRANZCR, Study Director — Gold Coast University Hospital; Laetitia E de Villiers MBCHB FRANZCR, Principal Investigator — Gold Coast University Hospital; Jason D Wenderoth BSc MBBS (Hons 1) FRANZCR, Principal Investigator — Prince of Wales Hospital; Albert Chiu MBBS (Hons.) FRANZCR, Principal Investigator — Sir Charles Gardiner Hospital; Nathan Manning BApSci, BSci(Hons) MBBS FRANZCR CCINR, Principal Investigator — Liverpool Hospital
Locations (4):
- Australia (4):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Sir Charles Gairdner Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the Australian Government Data Sharing Policy, the NHMRC Open Access Policy and the Clinical Trials Registration and Results Information Submission rule.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: To align with national recommendations for data sharing, the SCOPE-AUS metadata (description of the data) shall be published in a metadata record through Research Data Australia Registry, an entity of the Australian National Data Service. The goal is to ensure that data that is unique to the discipline of Interventional Neuroradiology is available for reuse in future research purposes.
  The SCOPE-AUS metadata will be available at 12 months following primary publication until 48 months.
Access Criteria: Access shall be conditional; re-users must be genuine researchers whose proposed use of the data has been approved by an Ethics committee. Re-users are required to cite the SCOPE-AUS dataset in any scholarly outputs. This proposed strategy will uphold Australian privacy laws. The Sponsor/Coordinating Principal Investigator/SCOPE-AUS research team will ultimately retain oversight of all future uses of the data.
URL: https://researchdata.ands.org.au/